CLINICAL TRIAL: NCT02092311
Title: Assessing Post-operative Rates of Recurrence, Hydrocele and Testicular Atrophy in Patients Operated With a New Approach of Varicocelectomy Named Combined Mini-incision Microscopic Varicocelectomy (CMMV)
Brief Title: Assessing the Rates of Major Complications in Combined Mini-incision Microscopic Varicocelectomy
Acronym: CMMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omid Fertility Center (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMMV
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Varicocele
Keywords: varicocele; varicocelectomy; complications of varicocelectomy; Recurrence of varicocele; Post-varicocelectomy testicular atrophy; Post-varicocelectomy hydrocele
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined Microscopic Varicocelectomy (Experimental): Patients in this arm were operated with Combined Mini-incision Microscopic approach
  Interventions: Procedure: Combined Microscopic Varicocelectomy
- Inguinal and Subinguinal Varicocelectomy (Active Comparator): Patients in this arm have the same including criteria as Experimental arm but they were operated with conventional and currently popular approach of Microscopic Inguinal and Sub inguinal varicocelectomy suggested by Goldstien and associates
  Interventions: Procedure: Inguinal and Subinguinal varicocelectomy

INTERVENTIONS:
Procedure: Combined Microscopic Varicocelectomy — After making a mini-incision at inguinal level, veins are evaluated, and if the including criteria (Complexity and tortuosity of the veins and/or existence of veins that are contiguous with arteries so that separating and ligation of the veins could jeopardize the artery) are existed, only external spermatic vein, if dilated, is ligated at the depth of the inguinal canal, and other veins are left alone for prevention of damage to the artery. Subsequently, another mini-incision is made at high inguinal level and the rest of surgery is conducted by retroperitoneal approach, which is also done microscopically
  Arms: Combined Microscopic Varicocelectomy
Procedure: Inguinal and Subinguinal varicocelectomy — Microscopic Inguinal and Sub inguinal varicocelectomy, recommended by Goldstein and associates, are currently popular approaches. In this approach the spermatic cord structures are pulled up and out of the wound so that the testicular artery, lymphatics, and small periarterial veins may be more easily identified. In addition, an inguinal or subinguinal approach allows access to external spermatic and even gubernacular veins.
  Arms: Inguinal and Subinguinal Varicocelectomy

SUMMARY:
The purpose of this study is to determine the rates of major post-varicocelectomy complications (Recurrence, Hydrocele and Testicular Atrophy) in patients operated with a new method named Combined Mini-incision Microscopic Varicocelectomy. The study hypothesis is that using this method will lead to less major complications of recurrence, hydrocele, and also less incidental injuries to the arteries that will result less testicular atrophy

DETAILED DESCRIPTION:
The sample is selected from the patients who were referred to our center for surgical treatment of varicocele. Most of them were diagnosed after being evaluated for infertility.

All of them were operated by a single experienced and expert microscopic surgeon.

Informed consent is received from all of the possible candidates in accordance to national and Declaration of Helsinki guidelines.

Selection of patients for undergoing Combined varicocelectomy was done during the operation due to the nature of including criteria.

In this method after making an incision at inguinal level, veins are evaluated and if the including criteria is existed, only external spermatic vein is ligated at the depth of the inguinal canal and other veins are left alone for prevention of damage to the artery. Then another mini incision is made at high inguinal level and the rest of surgery is conducted by retroperitoneal approach.

The incidence rate of major complications (recurrence, testicular atrophy, hydrocele) of experimental group is compared to the incidence rate of the same complications of the patients in control group that were operated with currently common inguinal and subinguinal microscopic varicocelectomy accompanied by testicular delivery, an approach that is suggested by Goldstein and associates.

The study hypothesis is that using this method will lead to less major complications including recurrence, hydrocele and also less incidental injuries to the arteries that will result to less testicular atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Complexity and tortuosity of the veins at inguinal level so that separating and ligation of the vein could lead to artery injury
* Veins which are contiguous with arteries so that separating and ligation of the vein could lead to artery injury

Exclusion Criteria:

* Prior surgery at inguinal level such as Herniorrhaphy, Orchiopexy,etc.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2006-01; Primary Completion 2013-09 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omid Pouyan, MD, Study Director — Omid Fertility Center; Navid Pooyan, MD, Principal Investigator — Omid Fertility Center; Robabeh Taheri Panah, MD, Study Chair — Infertility and Reproductive Health research center of Shahid Beheshti university of medical sciences; Ashraf Ale Yasin, MD, Study Chair — Omid Fertility Center; Marzieh Agha Hosseini, MD, Study Chair — Omid Fertility Center; Hojatollah Saeidi Saeid Abadi, P.H.D, Study Chair — Omid FC
Locations (1):
- Omid fertility center, Tehran, Tehran Province, Iran

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Microscopic Varicocelectomy: Combined Mini-Incision Microscopic Varicocelectomy
- Inguinal and Subinguinal Varicocelectomy: Patients in this arm have the same including criteria as Experimental arm but they were operated with conventional and currently popular approach of Microscopic Inguinal and Sub inguinal varicocelectomy suggested by Goldstien and associate
Period: Overall Study
Arm/Group | Combined Microscopic Varicocelectomy | Inguinal and Subinguinal Varicocelectomy
Started | 285 | 285
Completed | 285 | 285
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Combined Microscopic Varicocelectomy: Patients underwent Combined Mini-incision Microscopic Varicocelectomy
- Total: Total of all reporting groups
Arm/Group | Combined Microscopic Varicocelectomy | Inguinal and Subinguinal Varicocelectomy | Total
Number analyzed (Participants) | 285 | 285 | 570
Age, Continuous [Mean (Full Range); unit: years] | 31.2 [16 to 40] | 31.8 [22 to 39] | 31.5 [16 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 285 | 285 | 570
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 285 | 285 | 570

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Varicocele
Description: post-varicocelectomy recurrence is measured by physical exam at intervals of 10 days,3months and 6months after surgery
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Combined Microscopic Varicocelectomy | Inguinal and Subinguinal Varicocelectomy
Number analyzed (Participants) | 285 | 285
participants | 2 | 16

2. Secondary Outcome: Post-varicocelectomy Hydrocele
Description: Development of hydrocele is assessed by physical exam at intervals of 10 days,3months and 6months after surgery
Time Frame: 6months
Measure: Number; unit: Participants
Arm/Group | Combined Microscopic Varicocelectomy | Inguinal and Subinguinal Varicocelectomy
Number analyzed (Participants) | 285 | 285
Participants | 0 | 0

3. Other Pre Specified Outcome: Post-varicocelectomy Testicular Atrophy
Description: development of testicular atrophy is assessed by physical exam at intervals of 3 and 6 months after surgery
Time Frame: 6months
Measure: Number; unit: Participants
Arm/Group | Combined Microscopic Varicocelectomy | Inguinal and Subinguinal Varicocelectomy
Number analyzed (Participants) | 285 | 285
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Combined Microscopic Varicocelectomy | Inguinal and Subinguinal Varicocelectomy
Serious Adverse Events (participants affected / at risk) | 0/285 | 0/285
Other Adverse Events (participants affected / at risk) | 2/285 | 16/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Microscopic Varicocelectomy (N=285) | Inguinal and Subinguinal Varicocelectomy (N=285)
Testicular Atrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Microscopic Varicocelectomy (N=285) | Inguinal and Subinguinal Varicocelectomy (N=285)
Recurrent Varicocele (Reproductive system and breast disorders) | 2 | 16
Hydrocele (Reproductive system and breast disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No